CLINICAL TRIAL: NCT05905289
Title: Survival and Reproductive Outcomes After Fertility-sparing Surgery and Adjuvant Chemotherapy in Malignant Ovarian Germ Cell Tumors
Brief Title: Survival and Reproductive Outcomes of Malignant Ovarian Germ Cell Tumors
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mahmoud Ahmed Ismail Abd El Hameed, Principal Investigator, Cairo University
Other Study IDs: N-181-2023
Record Dates: First submitted 2023-06-07; First posted 2023-06-15 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Fertility Issues
Keywords: Ovarian germ cell tumors; Fertility sparing
MeSH Terms: conditions — Infertility | interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- group A: young female patients diagnosed with malignant ovarian germ cell tumors underwent fertility-sparing surgery and adjuvant chemotherapy will be retrospectively investigated
  Interventions: Other: observational study

INTERVENTIONS:
Other: observational study — no intervention as it is an observational study

SUMMARY:
Malignant ovarian germ cell tumor patients conducted fertility-sparing surgery and adjuvant chemotherapy in Kasr El-Aini Hospital - Faculty of Medicine - Cairo University from January 2012 to December 2016 will be retrospectively investigated.

DETAILED DESCRIPTION:
MOGCT patients conducted fertility-sparing surgery and adjuvant chemotherapy with complete follow up data, younger than 35 years old at first treatment, in Kasr El-Aini Hospital - Faculty of Medicine - Cairo University ( Department of Obstetrics & Gynecology and Center of Clinical Oncology and Nuclear Medicine ) from January 2012 to December 2016 will be retrospectively investigated.

Diagnosis of MOGCT was revealed by pelvic mass, abdominal pain, and elevated tumor markers like α-fetoprotein (AFP), human choionic gonadotophin (HCG) and lactate dehydrogenase (LDH) and confirmed by surgical procedure and pathological diagnosis. Pathological diagnosis was confirmed according to the 2014 World Health Organization classification of tumors of female reproductive organs. Tumors were staged according to American Joint Committee of Cancer (AJCC), TNM and FIGO staging system for Ovarian and Primary Peritoneal Cancer.

Fertility sparing surgery preserves uterus and the contralateral ovary with or without comprehensive staging (omentectomy and lymphadenectomy) by open laparotomy. Adjuvant chemotherapy was scheduled based on histopathology, grade and stage. All patients received chemotherapy, but with different schemes and courses The data including: subjects' demographics, clinical and pathological characteristics, treatment received, survival outcome and reproductive outcomes including pregnancy rate ( natural conception ) and live birth rate will be investigated. Follow-up data until January 31, 2022 will be collected from hospital records and telephone interview.

ELIGIBILITY:
Inclusion Criteria:

* Age : younger than 35 years old at first treatment.
* Fertility-sparing surgery and adjuvant chemotherapy.
* Pathological diagnosis of malignant ovarian germ cell tumor.

Exclusion Criteria:

* Patients with benign ovarian germ cell tumors e.g. mature teratoma.
* Concurrent malignancy.
* Severe comorbidities that may affect ovarian reproductive function.

Ages: 18 Years to 35 Years | Sex: Female
Age Groups: Adult
Study Population: Malignant ovarian germ cell tumor patients conducted fertility-sparing surgery and adjuvant chemotherapy with complete follow up data from January 2012 to December 2016 will be retrospectively investigated.
Sampling Method: Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2023-12-11 (Actual)

PRIMARY OUTCOMES:
reproductive outcomes | 5 years
  To report and analyze reproductive outcome including pregnancy rate and live birth rate after fertility-sparing surgery and adjuvant chemotherapy in malignant ovarian germ cell tumors

SECONDARY OUTCOMES:
Clinico-pathological characteristics of MOGCTs. | 5 years
  the clinical presentation and histopathological features of MOGCTs.

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Ahmed Abd El Hameed, MD, Principal Investigator — Kasr Al Ainy Hospital, Faculty of Medicine, Cairo University
Locations (1):
- Department of Obstetrics & Gynecology, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No